CLINICAL TRIAL: NCT01190059
Title: Normothermic Ex Vivo Lung Perfusion (EVLP) For An Improved Assessment of Donor Lungs For Transplantation
Acronym: HELP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: XVIVO Perfusion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VIT-001-TOR; 139150 (Other: Health Canada)
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Lung Transplantation
Keywords: Lung; Transplantation; Lung Transplantation; Transplantation Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EVLP Group (Experimental): EVLP Group are those recipient lung transplant patients that received donor lungs that had been placed on the ex vivo lung perfusion system with Steen Solution™ .
  Interventions: Drug: Ex vivo lung perfusion with Steen Solution™

INTERVENTIONS:
Drug: Ex vivo lung perfusion with Steen Solution™ — The circuit is primed with 2,000cc Steen Solution™. At one hour of EVLP, 500 cc of circulated perfusate was removed and replenished with 500 cc of fresh perfusate. After that, 250 cc of perfusate was exchanged every hour.

SUMMARY:
The use of ex vivo lung perfusion (EVLP) will allow for a secondary evaluation technique for donor lungs that fail to meet standard acceptability criteria. This advanced assessment might lead to increased utilization rates of donor lungs and improved outcomes after lung transplantation.

DETAILED DESCRIPTION:
Human donor lungs that do not meet the standard clinical criteria for donor lung utilization but fit into the study inclusion criteria will be retrieved from the donor using current donor lung retrieval techniques.

These lungs will be brought to the study transplant center to be re-assessed by the transplant team. The lungs will be physiologically assessed during ex vivo perfusion with Steen Solution. Perfusion of these lungs will be performed using Steen solution with the addition of methylprednisolone, heparin and antibiotics. With respect to the decision of lung utilization those organs with a delta pO2 (Δ pO2 = Pulmonary vein pO2 - pulmonary artery pO2) during ex vivo perfusion assessment > 350mmHg, good lung compliance, and a favorable opinion of the transplant surgeon will be considered transplantable. Lungs will be excluded for transplantation: if the Δ pO2 is less than 350mmHg or if they demonstrate >10% deterioration in any of the following functional parameters: pulmonary vascular resistance (PVR), dynamic compliance or airway pressures. Lungs will also be excluded if they are deemed unsuitable based on the clinical judgment of the lung transplant surgeon.

ELIGIBILITY:
Inclusion Criteria for donor lung:

1. Recipient to undergo a single or bilateral Lung Transplantation
2. Last donor PaO2/FiO2 ≤ 300mmHg
3. Poor oxygenation and/or poor lung compliance is the primary reason for unsuitability
4. Absence of pneumonia, persistent purulent secretion on bronchoscopy or significant mechanical trauma

Exclusion Criteria:

1. Infection
2. Aspiration
3. Significant mechanical lung injury - contusion
4. Infectious diseases : HIV, Hepatitis B and C, HTLV & Syphilis
5. Malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-08; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
PGD scores in the first 72 hours after lung transplantation. | 72 hours
  Immediate lung function is one of the key factors in determining the impact of donor lung quality, therefore the PGD score within 72 hrs was selected as the primary endpoint.
30 day Mortality | 30 days
  Mortality at 30 days post transplant

SECONDARY OUTCOMES:
Extra-corporeal membrane oxygenation use | 30 days
  If the patient needed to be placed on extra-corporeal membrane oxygenation after transplantation.
Bronchial complications | 30 days
  To see if there was an increased risk for bronchial complications
Ventilator duration | 30 days
  How long was the patient on the ventilator after lung transplantation and was there an increased time on ventilator for the patient after EVLP.
Intensive Care Unit length of stay | 30 days
Hospital length of stay | 30 days
  Time in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Shaf Keshavjee, MD,MSc,FRCSC, Principal Investigator — University of Toronto / Toronto General Hospital
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Pierre AF, Sekine Y, Hutcheon MA, Waddell TK, Keshavjee SH. Marginal donor lungs: a reassessment. J Thorac Cardiovasc Surg. 2002 Mar;123(3):421-7; discussion, 427-8. doi: 10.1067/mtc.2002.120345. PMID 11882811
- [Background] de Perrot M, Liu M, Waddell TK, Keshavjee S. Ischemia-reperfusion-induced lung injury. Am J Respir Crit Care Med. 2003 Feb 15;167(4):490-511. doi: 10.1164/rccm.200207-670SO. PMID 12588712
- [Background] Cypel M, Rubacha M, Yeung J, Hirayama S, Torbicki K, Madonik M, Fischer S, Hwang D, Pierre A, Waddell TK, de Perrot M, Liu M, Keshavjee S. Normothermic ex vivo perfusion prevents lung injury compared to extended cold preservation for transplantation. Am J Transplant. 2009 Oct;9(10):2262-9. doi: 10.1111/j.1600-6143.2009.02775.x. Epub 2009 Aug 6. PMID 19663886
- [Background] D.M. Karamanou, H.R. Walden, S. Bean, et al. The Effect of Ex-Vivo Perfusion on the Inflammatory Profile of the Donor Lung. J Heart Lung Transplant 2010:Vol. 29, Issue 2, Supplement, Page S165.
- [Background] Inci I, Ampollini L, Arni S, Jungraithmayr W, Inci D, Hillinger S, Leskosek B, Vogt P, Weder W. Ex vivo reconditioning of marginal donor lungs injured by acid aspiration. J Heart Lung Transplant. 2008 Nov;27(11):1229-36. doi: 10.1016/j.healun.2008.07.027. Epub 2008 Oct 1. PMID 18971096
- [Background] Steen S, Sjoberg T, Pierre L, Liao Q, Eriksson L, Algotsson L. Transplantation of lungs from a non-heart-beating donor. Lancet. 2001 Mar 17;357(9259):825-9. doi: 10.1016/S0140-6736(00)04195-7. PMID 11265950
- [Background] Ingemansson R, Eyjolfsson A, Mared L, Pierre L, Algotsson L, Ekmehag B, Gustafsson R, Johnsson P, Koul B, Lindstedt S, Luhrs C, Sjoberg T, Steen S. Clinical transplantation of initially rejected donor lungs after reconditioning ex vivo. Ann Thorac Surg. 2009 Jan;87(1):255-60. doi: 10.1016/j.athoracsur.2008.09.049. PMID 19101308
- [Background] Steen S, Ingemansson R, Eriksson L, Pierre L, Algotsson L, Wierup P, Liao Q, Eyjolfsson A, Gustafsson R, Sjoberg T. First human transplantation of a nonacceptable donor lung after reconditioning ex vivo. Ann Thorac Surg. 2007 Jun;83(6):2191-4. doi: 10.1016/j.athoracsur.2007.01.033. PMID 17532422
- [Derived] Cypel M, Yeung JC, Liu M, Anraku M, Chen F, Karolak W, Sato M, Laratta J, Azad S, Madonik M, Chow CW, Chaparro C, Hutcheon M, Singer LG, Slutsky AS, Yasufuku K, de Perrot M, Pierre AF, Waddell TK, Keshavjee S. Normothermic ex vivo lung perfusion in clinical lung transplantation. N Engl J Med. 2011 Apr 14;364(15):1431-40. doi: 10.1056/NEJMoa1014597. PMID 21488765